CLINICAL TRIAL: NCT03444636
Title: The Efficacy and Safety of Multimodal Analgesia in Children and Adolescents After the Ravitch Procedure and Thoracotomy - a Prospective Randomized Study
Brief Title: Multimodal Analgesia in Children and Adolescents After the Ravitch Procedure and Thoracotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute for Tuberculosis and Lung Diseases, Poland (Other)
Responsible Party: Principal Investigator, Lucyna Tomaszek, PhD, RN, Director of Nursing, Specialist Nurse in Anesthesia and Intensive Care, National Institute for Tuberculosis and Lung Diseases, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10.7
Record Dates: First submitted 2018-02-16; First posted 2018-02-23 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pain, Postoperative; Surgery, Thoracic
Keywords: Multimodal analgesia; Thoracic epidural; Postoperative pain; Postoperative Complications; Patient Satisfaction
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Patient Satisfaction | interventions — Ropivacaine; Fentanyl; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine/Fentanyl (Experimental)
  Interventions: Drug: Ropivacaine/Fentanyl
- Bupivacaine/Fentanyl (Active Comparator)
  Interventions: Drug: Bupivacaine/Fentanyl

INTERVENTIONS:
Drug: Ropivacaine/Fentanyl — Ropivacaine 0.2% with Fentanyl 5 µg/ml; flow rate of 0.1 ml/kg/hr
  Other Names: ROPIVACAINE HYDROCHLORIDE 10 mg/ml
  Arms: Ropivacaine/Fentanyl
Drug: Bupivacaine/Fentanyl — Bupivacaine 0.125% with Fentanyl 5 µg/ml; flow rate of 0.1 ml/kg/hr
  Other Names: BUPIVACAINE HYDROCHLORIDE 0.5%
  Arms: Bupivacaine/Fentanyl

SUMMARY:
The study was performed in patients aged 6-18 years after the Ravitch procedure and thoracotomy. The primary aim of the study was to evaluate the efficacy and safety of pain control provided by the multimodal approach that involves the continuous infusion ropivacaine with fentanyl vs. bupivacaine with fentanyl through thoracic epidural catheter. Secondary aims were to identify the determinants of acute post-operative pain at rest, during deep breathing and coughing.

DETAILED DESCRIPTION:
The subjects were randomized to the Ropivacaine/Fentanyl (RF) or Bupivacaine/Fentanyl (BF) group.

To perform a thoracic surgical procedure, all patients were premedicated with midazolam, and then, paracetamol, non-steroidal anti-inflammatory drugs, fentanyl, propofol, pancuronium or rocuronium (in children < 10 years old) and suprane were used to introduce and maintain the anesthesia. Thoracic epidural catheters were placed following induction of anesthesia and endotracheal intubation.

Intraoperative analgesia was introduced by a single dose of lidocaine 2% (2 mg/kg). Then after 15 minutes, the patients from the RF group received ropivacaine 1% (1-3 mg/kg) and those from the BF group bupivacaine 0.5% (0.5-1 mg/kg). After 60 minutes 0.2% ropivacaine solution with fentanyl or 0.125% solution of bupivacaine with fentanyl was infused with the flow rate of 0.1 ml/kg/hr.

Depending on the allocation to the group, postoperative analgesia was continued either with 0.2% ropivacaine and fentanyl or 0.125% bupivacaine and fentanyl, based on the concentration and the flow rate described above. In addition, intravenous paracetamol was administered as standard every 6 hours (the maximum of 60 mg/kg daily) along with non steroidal anti-inflammatory drugs. In children > 14 years of age, ketoprofen was injected at the dose of 1 mg/kg (the maximum of 200 mg daily) and in younger children ibuprofen (orally or rectally, up to 30 mg/kg daily) every 8 hours. Metamizol was given as a "rescue drug" (20 mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Elective thoracic surgery (thoracotomy or Ravitch procedure);
* Analgesia: continuous thoracic epidural analgesia.

Exclusion Criteria:

* American Society of Anesthesiologists physical status >III;
* History of chronic pain or preoperative opioid use;
* Oncological treatment;
* Impaired verbal communication;
* Removal of epidural catheter <24 h postoperatively;
* Lack of postoperative chest drainage.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 2015-03-02 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity scores at rest (FLACC for patients <7 y.o., Numerical Rating Scale for patients >7 y.o.) | postoperative day: 0-3
Pain intensity scores during deep breathing (FLACC for patients <7 y.o., Numerical Rating Scale for patients >7 y.o.) | postoperative day: 0-3
Pain intensity scores during coughing (FLACC for patients <7 y.o., Numerical Rating Scale for patients >7 y.o.) | postoperative day: 0-3
Side Effect Occurrence | first 3 days after surgery

SECONDARY OUTCOMES:
Total fentanyl consumption [µg] | postoperative day: 0-3
The number of doses of metamizol as a "rescue drug" | postoperative day: 0-3
The number of nursing interventions undertaken to relive pain > 2/10 pts | postoperative day: 0-3
Patient satisfaction | postoperative day 3
  Satisfaction was evaluated on a 4-item scale: analgesia was rated as insufficient, poor, good or very good.

CONTACTS AND LOCATIONS:
Overall Officials: Lucyna Tomaszek, PhD, Study Director — National Institute for Tuberculosis and Lung Diseases, Poland
Locations (1):
- Institute for Tuberculosis and Lung Diseases, Pediatric Division, Rabka-Zdrój, Małopolska, Poland

REFERENCES:
- [Background] Misiolek H, Cettler M, Woron J, Wordliczek J, Dobrogowski J, Mayzner-Zawadzka E. The 2014 guidelines for post-operative pain management. Anaesthesiol Intensive Ther. 2014 Sep-Oct;46(4):221-44. doi: 10.5603/AIT.2014.0041. No abstract available. PMID 25293474
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Schnabel A, Thyssen NM, Goeters C, Zheng H, Zahn PK, Van Aken H, Pogatzki-Zahn EM. Age- and procedure-specific differences of epidural analgesia in children--a database analysis. Pain Med. 2015 Mar;16(3):544-53. doi: 10.1111/pme.12633. Epub 2015 Jan 19. PMID 25599577
- [Background] Ecoffey C, Lacroix F, Giaufre E, Orliaguet G, Courreges P; Association des Anesthesistes Reanimateurs Pediatriques d'Expression Francaise (ADARPEF). Epidemiology and morbidity of regional anesthesia in children: a follow-up one-year prospective survey of the French-Language Society of Paediatric Anaesthesiologists (ADARPEF). Paediatr Anaesth. 2010 Dec;20(12):1061-9. doi: 10.1111/j.1460-9592.2010.03448.x. PMID 21199114
- [Background] Lejus C, Surbled M, Schwoerer D, Renaudin M, Guillaud C, Berard L, Pinaud M. Postoperative epidural analgesia with bupivacaine and fentanyl: hourly pain assessment in 348 paediatric cases. Paediatr Anaesth. 2001 May;11(3):327-32. doi: 10.1046/j.1460-9592.2001.00659.x. PMID 11359592
- [Background] Tomaszek L, Fenikowski D, Komotajtys H, Gawron D. Ropivacaine/Fentanyl vs. Bupivacaine/Fentanyl for Pain Control in Children after Thoracic Surgery: A Randomized Study. Pain Manag Nurs. 2019 Aug;20(4):390-397. doi: 10.1016/j.pmn.2019.02.007. Epub 2019 May 15. PMID 31103498
- [Background] Tomaszek L, Fenikowski D, Gawron D, Komotajtys H. Comparative efficacy of continuous infusion of bupivacaine/fentanyl and ropivacaine/fentanyl for paediatric pain control after the Ravitch procedure and thoracotomy. A prospective randomized study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2019 Dec;163(4):366-373. doi: 10.5507/bp.2018.072. Epub 2018 Nov 16. PMID 30451243